CLINICAL TRIAL: NCT02686749
Title: Catheter Ablation vs. Medical Therapy in Congested Hearts With AF (CATCH-AF in Patients With Impaired LV Function): An Early Ablation Strategy Study Impact on Health Care Utilization
Brief Title: Catheter Ablation vs. Medical Therapy in Congested Hearts With AF
Acronym: CATCH-AF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: unable to reach enrollment goal
Sponsor: The Cleveland Clinic (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bio-858981
Record Dates: First submitted 2016-02-05; First posted 2016-02-19 (Estimated); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Congestive Heart Failure; Left Ventricular Failure; Atrial Fibrillation
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Study randomizes subjects to already FDA approved treatment modalities. Approved anti-arrhythmic medications or AF ablation. There are no investigational drug or devices used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- AF catheter Ablation (Active Comparator): Pulmonary Vein Isolation catheter ablation for treatment of AF. AF catheter ablation is an FDA approved treatment for AF
  Interventions: Device: Catheter Ablation
- FDA approved anti arrhythmic drug (Active Comparator): FDA approved anti arrhythmic drug for the treatment of AF will be based on treating physicians' preference in accordance to guidelines.
  Interventions: Drug: FDA approved anti arrhythmic drug

INTERVENTIONS:
Device: Catheter Ablation — During ablation, a doctor inserts a catheter through blood vessels into the heart. The doctor looks at the electrical activity of the heart. The catheter is used to determine which areas of the heart are causing AF. After the area is identified, the doctor uses a special machine delivers energy through the catheter to tiny areas of the heart muscle that is causing AF. This energy causes a scar in the tissue which "disconnects" the pathway of the AF.
  Other Names: Pulmonary Vein Isolation
  Arms: AF catheter Ablation
Drug: FDA approved anti arrhythmic drug — Anti arrhythmic drug medical treatment will be based on treating physicians discretion following standard clinical guidelines
  Arms: FDA approved anti arrhythmic drug

SUMMARY:
This study is a multi-center, randomized, unblinded, clinical trial. The objective is to determine if catheter-based atrial fibrillation (AF) ablation is superior to medical treatment in patients with impaired left ventricular (LV) function who have been diagnosed with symptomatic AF within the past 12 months.

DETAILED DESCRIPTION:
The purpose of the trial is to compare two different approved treatments for recently diagnosed AF: anti-arrhythmic medications and AF ablation. The study will be conducted to determine if one treatment is more effective than the other for patients with AF and heart failure. About 220 subjects with newly diagnosed AF from hospitals in the United States will take part in this study. Subjects will be randomized in a 1:1 fashion to either AF catheter ablation or anti-arrhythmic medication for treatment of AF. Both therapies are considered Standard of Care.

ELIGIBILITY:
Inclusion Criteria:

* must be 18 years of age or older
* Provide signed written Informed Consent
* symptomatic AF documented by EKG or heart rhythm monitoring within 12 months
* patients should be on optimal medical therapy for heart failure for 3 months prior to randomization. Adjustments to medications within this 3 month period are permitted.
* chronically impaired LV function defined as EF between 20%-45% within last 3 months
* all patients should be on an optimal therapy for impaired LV function
* ability to complete 6 minute walk test
* eligible for catheter ablation and anti-arrhythmic drugs

Exclusion Criteria:

* women of childbearing potential unless post- menopausal or surgically sterile
* patients hospitalized for heart failure within the 3 months prior to randomization
* reversible causes of AF such as pericarditis, thyroid disorders, acute alcohol intoxication, recent major surgical procedures or trauma
* recent reversible LV impairment that may be attributed to AF with rapid ventricular response and may improve with introduction of rate control
* valvular heart disease requiring surgical intervention
* Coronary Artery Disease (CAD) requiring surgical or percutaneous intervention
* early post-operative AF (within 3 months of surgery)
* previous MAZE or left atrial instrumentation (including ablation and left atrial appendage exclusion)
* history of Atrioventricular Node (AVN) ablation
* hypertrophic cardiomyopathy
* prolonged QT interval
* liver failure
* renal failure requiring dialysis
* social factors that would preclude follow up or make compliance difficult- history of drug, alcohol or substance abuse
* contraindications to the use of AADs and/or anticoagulation therapy
* Currently enrolled in, or discontinued within the last 30 days from a clinical trial involving an investigational product or non-approved use of a drug or device or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* severe pulmonary disease
* documented intra-atrial thrombus, tumor, or structural abnormality which precludes catheter introduction
* unwilling to comply with protocol requirements or deemed by the investigator to be unfit for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oussama Wazni, MD, Principal Investigator — The Cleveland Clinic
Locations (6):
- United States (6):
  - Hartford Hospital, Hartford, Connecticut
  - Cleveland Clinic Akron General, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kannel WB, Abbott RD, Savage DD, McNamara PM. Epidemiologic features of chronic atrial fibrillation: the Framingham study. N Engl J Med. 1982 Apr 29;306(17):1018-22. doi: 10.1056/NEJM198204293061703. PMID 7062992
- [Background] Van den Berg MP, Tuinenburg AE, Crijns HJ, Van Gelder IC, Gosselink AT, Lie KI. Heart failure and atrial fibrillation: current concepts and controversies. Heart. 1997 Apr;77(4):309-13. doi: 10.1136/hrt.77.4.309. PMID 9155607
- [Background] Chen MS, Marrouche NF, Khaykin Y, Gillinov AM, Wazni O, Martin DO, Rossillo A, Verma A, Cummings J, Erciyes D, Saad E, Bhargava M, Bash D, Schweikert R, Burkhardt D, Williams-Andrews M, Perez-Lugones A, Abdul-Karim A, Saliba W, Natale A. Pulmonary vein isolation for the treatment of atrial fibrillation in patients with impaired systolic function. J Am Coll Cardiol. 2004 Mar 17;43(6):1004-9. doi: 10.1016/j.jacc.2003.09.056. PMID 15028358
- [Background] Wyse DG. Some recent randomized clinical trials in the management of atrial fibrillation. J Interv Card Electrophysiol. 2003 Oct;9(2):223-8. doi: 10.1023/a:1026292609252. PMID 14574035
- [Background] Corley SD, Epstein AE, DiMarco JP, Domanski MJ, Geller N, Greene HL, Josephson RA, Kellen JC, Klein RC, Krahn AD, Mickel M, Mitchell LB, Nelson JD, Rosenberg Y, Schron E, Shemanski L, Waldo AL, Wyse DG; AFFIRM Investigators. Relationships between sinus rhythm, treatment, and survival in the Atrial Fibrillation Follow-Up Investigation of Rhythm Management (AFFIRM) Study. Circulation. 2004 Mar 30;109(12):1509-13. doi: 10.1161/01.CIR.0000121736.16643.11. Epub 2004 Mar 8. PMID 15007003

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AF Catheter Ablation | FDA Approved Anti Arrhythmic Drug
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — terminated for poor enrollment | 2 | 2

BASELINE CHARACTERISTICS:
Population: Trial terminated due to poor enrollment and no analysis was performed. No subjects completed study. Did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results.
Groups:
- Total: Total of all reporting groups
Arm/Group | AF Catheter Ablation | FDA Approved Anti Arrhythmic Drug | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants] — Population: Trial terminated due to poor enrollment. No subjects completed study. Did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 2 | 0 | 2
    >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Trial terminated due to poor enrollment. No subjects completed study. No data analyzed. Did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results. Population: Trial terminated due to poor enrollment. No subjects completed study. No data analyzed. Did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Trial terminated due to poor enrollment. No subjects completed study. No data analyzed. Did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results. Population: Trial terminated due to poor enrollment. No subjects completed study. No data analyzed. Did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results.

OUTCOME MEASURES:

1. Primary Outcome: First Hospitalization for Heart Failure, Recurrence of AF or Direct Current Cardioversion
Description: Time measured in days to first hospitalization for heart failure, recurrence of AF or Direct Current cardioversion after the treatment period (first 3 months post enrollment or post procedure during which repeat ablation can be performed and titration of AADs can be performed).
Time Frame: 12 months
Population: Trial terminated due to poor enrollment. No subjects completed study. Did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results.
Arm/Group | AF Catheter Ablation | FDA Approved Anti Arrhythmic Drug
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Total Number of Cardiovascular Hospitalization
Description: total number of cardiovascular hospitalization measured by hospitalization admissions
Time Frame: 15 months
Population: as for outcome 1
Arm/Group | AF Catheter Ablation | FDA Approved Anti Arrhythmic Drug
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Recurrence if AF Lasting Longer Than 30 Seconds
Description: time measured in days to recurrence of AF lasting longer than 30 seconds
Time Frame: 15 months
Population: as for outcome 1
Arm/Group | AF Catheter Ablation | FDA Approved Anti Arrhythmic Drug
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Distance Walked in a 6-mile Walk Test
Description: change in distance walked in 6 mile walk test
Time Frame: 3 months through 15 months
Population: as for outcome 1
Arm/Group | AF Catheter Ablation | FDA Approved Anti Arrhythmic Drug
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in the Rand 36-Item Health Survey
Description: change in the Rand 36-Item Health Survey reflective of change in patient's quality of life
Time Frame: 3 months through 15 months
Population: as for outcome 1
Arm/Group | FDA Approved Anti Arrhythmic Drug | AF Catheter Ablation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Ejection Fraction (EF)
Description: Change in Ejection Fraction heart failure measurement (percentage)
Time Frame: baseline through15 months
Population: as for outcome 1
Arm/Group | AF Catheter Ablation | FDA Approved Anti Arrhythmic Drug
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Trial was terminated before the outcome measure data were collected.
Arm/Group | AF Catheter Ablation | FDA Approved Anti Arrhythmic Drug
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Trial terminated due to poor enrollment. No subjects completed study. Did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT02686749/Prot_SAP_000.pdf